CLINICAL TRIAL: NCT00063154
Title: A Phase II, Open-label, Multicenter Study to Evaluate the Effect of Tumor-based HER2 Activation on the Efficacy of rhuMAb 2C4 (Pertuzumab) in Subjects With Recurrent Non-Small Cell Lung Cancer
Brief Title: Safety and Effect of Pertuzumab in Patients With Advanced Non-Small Cell Lung Cancer, Which Has Progressed After Prior Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC2572g; NCT00095602 (obsolete NCT alias)
Record Dates: First submitted 2003-06-20; First posted 2003-06-25 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pertuzumab (Experimental): Participants received pertuzumab intravenously on Day 1 of every 3 week cycle for up to 1 year (up to 17 treatment cycles). Subjects received pertuzumab at a loading dose of 840 mg in Cycle 1 followed by a dose of 420 mg in Cycles 2 and beyond.
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — Pertuzumab was supplied as a single-use liquid formulation.

SUMMARY:
The purpose of this study is to determine if the study drug pertuzumab is effective in treating patients with advanced lung cancer that has recurred following prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Tumor accessible to biopsy and willingness to undergo tumor biopsy
* Age >= 18 years
* Recurrent, histologically documented NSCLC, i.e., squamous cell, adeno-, or large cell anaplastic carcinoma. A cytologic diagnosis is acceptable (i.e. fine-needle aspiration or pleural fluid cytology).
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension (bilateral dimensions should be recorded). Each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain X-ray, CT, and MRI, or >= 10 mm when measured by spiral CT.
* Progression of disease during, or after completion of, at least one prior chemotherapy regimen, which should have contained either a platinum, a taxane or a vinca alkaloid (e.g. vinorelbine). There is no upper limit on the number of prior chemotherapy regimens each subject may have received.
* Recovery from reversible acute effects of prior chemotherapy regimens or radiotherapy to NCI-CTC Grade <= 1 (excluding alopecia)
* ECOG performance status of 0 or 1
* Use of an effective means of contraception for men, or for women of childbearing potential
* Absolute neutrophil count >= 1500/mL, platelet count of >= 75,000/mL and hemoglobin >= 9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbepoetin [Aranesp] is permitted)
* Serum bilirubin <= 1.5 x the upper limit of normal (ULN) and alkaline phosphatase, AST, and ALT <= 2.5 x ULN (ALT, AST, and alkaline phosphatase <= 5 x ULN for subjects with liver metastases)
* Serum creatinine <= 1.5 x ULN
* Internalized normalized ratio (INR) < 1.5 and activated partial thromboplastin time (aPTT) < 1.5 ULN (except for subjects receiving warfarin)

Exclusion Criteria:

* Prior treatment with any HER pathway inhibitors (e.g., Herceptin [Trastuzumab], Iressa [gefitinib], Tarceva [erlotinib hydrochloride], C225, CI1033, TAK165
* Treatment with other experimental anti-cancer agents within 4 weeks prior to Day 1
* Histologically documented bronchioalveolar carcinoma
* History or clinical or radiographic evidence of central nervous system or brain metastases
* Ejection fraction, determined by ECHO, <50%
* Uncontrolled hypercalcemia (> 11.5 mg/dL)
* Prior exposure of > 360 mg/m2 doxorubicin or liposomal doxorubicin, > 120 mg/m2 mitoxantrone, or > 90 mg/m2 idarubicin
* Ongoing corticosteroid treatment, except for subjects who are on stable doses of < 20 mg of prednisone daily (or equivalent), or for subjects who are taking corticosteroids for non-malignant conditions
* History of other malignancies within 5 years of Day 1 except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, or basal or squamous cell skin cancer
* History of serious systemic disease, uncontrolled hypertension (diastolic blood pressure > 100 mmHg on two consecutive occasions), unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation, paroxysmal supraventricular tachycardia, or controlled hypertension are eligible)
* Ongoing liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Active infection requiring IV antibiotics
* Known human immunodeficiency virus infection
* Pregnancy or lactation
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1, with the exception of tumor biopsy for the purposes of the study
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-07; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Arizona Cancer Center, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial-Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pertuzumab
Started | 51
Completed | 0
Not Completed | 51
Not completed — Disease progression | 27
Not completed — Adverse Event | 2
Not completed — Physician Decision | 10
Not completed — Death | 3
Not completed — Reason unspecified | 1
Not completed — Did not receive treatment | 8

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who received any amount of pertuzumab.
Arm/Group | Pertuzumab
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)
Description: A best overall response could occur at any time during the study and was determined by Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target lesions (TL) or the disappearance of all non-TLs and normalization of tumor marker level. A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD. SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since the treatment started for TLs and the persistence of 1 or more non-TL(s) and/or the maintenance of tumor marker level above normal limits. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started or the appearance of one or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: Efficacy-evaluable population: Participants who received at least 2 doses of pertuzumab and either underwent at least 1 post-baseline assessment of response or died as a result of disease progression before any evaluation of response.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 35
percentage of participants
  Complete response | 0.0
  Partial response | 0.0
  Stable disease | 51.4
  Progressive disease | 48.6

2. Secondary Outcome: Number of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) With HER2 Phosphorylation + or - Tumors
Description: as for outcome 1
Time Frame: Baseline to the end of the study (up to 1 year)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 38
participants
  Complete response pHER2+ (n=4) | 0
  Partial response pHER2+ (n=4) | 0
  Stable disease pHER2+ (n=4) | 2
  Progressive disease pHER2+ (n=4) | 1
  No tumor assessment pHER2+ (n=4) | 1
  Unable to evaluate response pHER2+ (n=4) | 0
  Complete response pHER2- (n=34) | 0
  Partial response pHER2- (n=34) | 0
  Stable disease pHER2- (n=34) | 15
  Progressive disease pHER2- (n=34) | 13
  No tumor assessment pHER2- (n=34) | 5
  Unable to evaluate response pHER2- (n=34) | 1

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first day of pertuzumab treatment (Cycle 1, Day 1) to the time of documented disease progression (per RECIST) or death, whichever occurred first.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab
Number analyzed (Participants) | 35
weeks | 6.6 [6.0 to 14.7]

4. Secondary Outcome: Number of Participants Free From Disease Progression at 3, 6, and 12 Months
Description: Disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to the end of the study (up to 1 year)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 35
participants
  3 months | 8
  6 months | 1
  9 months | 0

ADVERSE EVENTS:
Description: Safety population: All participants who received any amount of pertuzumab.
Arm/Group | Pertuzumab
Serious Adverse Events (participants affected / at risk) | 15/43
Other Adverse Events (participants affected / at risk) | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab (N=43)
PNEUMONIA (Infections and infestations) | 7
CELLULITIS (Infections and infestations) | 1
SEPSIS (Infections and infestations) | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PAIN (General disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab (N=43)
DIARRHOEA (Gastrointestinal disorders) | 15
NAUSEA (Gastrointestinal disorders) | 8
VOMITING (Gastrointestinal disorders) | 5
CONSTIPATION (Gastrointestinal disorders) | 4
STOMATITIS (Gastrointestinal disorders) | 4
FATIGUE (General disorders) | 16
PAIN (General disorders) | 6
PYREXIA (General disorders) | 4
ASTHENIA (General disorders) | 3
CHILLS (General disorders) | 3
OEDEMA PERIPHERAL (General disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
ANXIETY (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 3
ANOREXIA (Metabolism and nutrition disorders) | 8
HEADACHE (Nervous system disorders) | 5
DIZZINESS (Nervous system disorders) | 3
RASH (Skin and subcutaneous tissue disorders) | 5
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3
ANAEMIA (Blood and lymphatic system disorders) | 3
EJECTION FRACTION DECREASED (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.